CLINICAL TRIAL: NCT04686565
Title: Evaluation The Effect of The Covid-19 Pandemic on Children With CerebralPalsy and The Caregivers' Quality of Life
Brief Title: Covid-19 Pandemic and Cerebral Palsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Damla Cankurtaran, Medical doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: CP-covid
Record Dates: First submitted 2020-12-23; First posted 2020-12-28 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Palsy; Covid19; Telemedicine; Caregiver Quality of Life; Disability, Developmental
MeSH Terms: conditions — Cerebral Palsy; COVID-19; Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigator aimed to analyzed the effect of Covid-19 pandemic on the physical-psychosocial and cognitive state of the children, to benefit form the health, education services and the caregiver's quality of life with telemedicine.

DETAILED DESCRIPTION:
Telemedicine is an application that provides remote healthcare services. Telemedicine method has been reported to be useful in chronic conditions such as cerebral palsy (CP). Patients with CP need regular follow-up, regular physiotherapy, orthosis use, using of antispasmodic drugs, repeated botulinum toxin applications or intrathecal baclofen to reduce spasticity and increase functionality. During the Covid-19 pandemic period, these patients could not come to their controls due to reasons such as difficulty in reaching the doctor, fear of infection transmission, could not continue physiotherapy, repeated botulinum toxin applications could not be performed and necessary operations could not be performed. In this cross sectional study, investigator aimed to analyzed the effect of Covid-19 pandemic on the physical-psychosocial and cognitive state of the children, to benefit form the health, education services and the caregiver's quality of life with telemedicine.

ELIGIBILITY:
Inclusion Criteria:

* Patients' ages between 3-18 years
* Caregiver of Patients diagnosed as Cerebral palsy
* Patients with routine follow-ups in our clinic
* Caregivers can be reach by phone

Exclusion Criteria:

* Patients' ages under 3 and over 18 years

  --Caregivers cannot be reach by phone
* Caregivers without quality of life results for the pre-pandemic period

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients between the ages of 3-18 who are followed up with a diagnosis of cerebral palsy in our clinic and their primary caregivers will be included
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
The status of the child to benefit from health-education services | 10 seconds
  With the 14-question questionnaire prepared by the authors, the reasons such as whether there is a disruption in the control of the patients, the reason for the flow, the use of oral medications, the use of orthoses, the application of botulinum toxin, if they are applied, the development of side effects, and the obstacle to distance education will be questioned.
Physical-psychosocial and cognitive state of the child | 10 seconds
  With five questions prepared by the investigators themselves, primary caregivers will be asked to evaluate their children's disease status, mobility level, spasticity, range of motion, communication and emotional state as better, the same or worse compared to the pre-pandemic period.
Caregivers' quality of life | 30 seconds
  The quality of life of the primary caregivers of the patients during the Covid-19 period will be evaluated with the Short Form-12 using the phone and compared with the results recorded in their pre-pandemic files.
  It is an abbreviation of 12 questions of the 8-item, 36-question short form -36 developed to evaluate the positive and negative aspects of the health status. Patients are asked to be evaluated considering the last four weeks. The total score ranges from 0 to 100 and higher scores indicate better quality of life
the Covid-19 fear levels of Caregivers | 10 seconds
  Fear of Covid-19 scale is being used to evaluated the Covid-19 fear levels of Caregivers by telephone.It is a 7-question questionnaire evaluating the fear associated with covid-19, which is evaluated with a five-item Likert scale. The lowest score is 7, the highest score is 35. As the score increases, the level of fear due to Covid-19 increases. Turkish validity and reliability has been made.

CONTACTS AND LOCATIONS:
Overall Officials: Damla Cankurtaran, MD, Principal Investigator — Diskapi Yildirim Beyazit Education and Research Hospital; Ece uNLU aKYUZ, Assoc Prof., Study Director — Diskapi Yildirim Beyazit Education and Research Hospital; Nihal Tezel, MD, Study Chair — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- Diskapi Education and Research Hospital, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ben-Pazi H, Beni-Adani L, Lamdan R. Accelerating Telemedicine for Cerebral Palsy During the COVID-19 Pandemic and Beyond. Front Neurol. 2020 Jun 26;11:746. doi: 10.3389/fneur.2020.00746. eCollection 2020. PMID 32670193
- [Background] Cacioppo M, Bouvier S, Bailly R, Houx L, Lempereur M, Mensah-Gourmel J, Kandalaft C, Varengue R, Chatelin A, Vagnoni J, Vuillerot C, Gautheron V, Dinomais M, Dheilly E, Brochard S, Pons C; ECHO Group. Emerging health challenges for children with physical disabilities and their parents during the COVID-19 pandemic: The ECHO French survey. Ann Phys Rehabil Med. 2021 May;64(3):101429. doi: 10.1016/j.rehab.2020.08.001. Epub 2020 Aug 18. PMID 32818674
- [Background] Satici B, Gocet-Tekin E, Deniz ME, Satici SA. Adaptation of the Fear of COVID-19 Scale: Its Association with Psychological Distress and Life Satisfaction in Turkey. Int J Ment Health Addict. 2021;19(6):1980-1988. doi: 10.1007/s11469-020-00294-0. Epub 2020 May 8. PMID 32395095